CLINICAL TRIAL: NCT05762029
Title: Treatment of Extracorporeal Membrane Oxygenation in Severe Poisoning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: poison ECMO
Record Dates: First submitted 2023-02-13; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-12

CONDITIONS: Poison;Medicinal; Extracorporeal Membrane Oxygenation
Keywords: Severe poisoning; Extracorporeal Membrane Oxygenation; Emergency medical care
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Due to respiratory and circulatory failure caused by acute server poisoning, patients accepting extracorporeal membrane oxygenation for treatment.

SUMMARY:
This is a prospective, multicentre clinical study to determine the value of the Extracorporeal Membrane Oxygenation in the treatment of critically ill poisoning patients and whether there are significant differences in the prognosis of different types or doses of poison/drug poisoning. These conclusions may guide us on how to correctly perform Extracorporeal Membrane Oxygenation, including whether or when should this treatment enabled, the mode of Extracorporeal Membrane Oxygenation, whether to combine blood purification, treatment schedule and disembarkation time.

DETAILED DESCRIPTION:
This study will be conducted in the Affiliated Hospital of Nantong University, the Sixth People's Hospital of Nantong University, the Branch of Affiliated Hospital of Nantong University, the People's Hospital of Qidong City, the People's Hospital of Rudong County, the People's Hospital of Rugao City, and the People's Hospital of Hai 'an City. It is expected that 60 patients with poisoning will be included, and the blood and urine samples of 60 patients will be collected and stored in the clinical trial sample database to evaluate and record the relevant indicators of the subjects. The relevant medical records in clinical treatment were analyzed and studied. Each subject will be numbered and a separate medical record will be established.

The purpose of this prospective multicenter observational clinical study was to 1) investigate the value of Extracorporeal Membrane Oxygenation in the treatment of fatal poisoning; 2) To investigate the changes of patients' organ functions (heart, lung, liver, kidney, brain) during the Extracorporeal Membrane Oxygenation operation and the influence on the removal of toxins. In order to obtain a more powerful clinical basis to guide the rational use of the Extracorporeal Membrane Oxygenation technology in patients with fatal poisoning.

ELIGIBILITY:
Inclusion Criteria:

* Severe intoxication resulting in cardiac arrest, refractory malignant arrhythmia, refractory shock, refractory heart failure, respiratory failure.
* Denying other available methods.
* Indications for the use of the Extracorporeal membrane oxygenation exist.

Exclusion Criteria:

* Severely impaired state of consciousness prior to cardiac arrest;
* Multiple organ dysfunction;
* Uncontrolled traumatic bleeding, massive gastrointestinal bleeding, and active intracranial hemorrhage;
* Left ventricular thrombosis; Severe aortic insufficiency.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe intoxication resulting in cardiac arrest, refractory malignant arrhythmia, refractory shock, refractory heart failure, respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2025-11-26 (Estimated)

PRIMARY OUTCOMES:
Death rate | through study completion, assessed up to 3 year
  Death rate is used to assess the treatment capacity of Extracorporeal membrane oxygenation.
Complication | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 days
  Complication is used to assess the side effects of Extracorporeal membrane oxygenation.
Partial pressure of oxygen | random time before performing extracorporeal membrane oxygenation
  PO₂ is used to indicate the state of internal respiration.
Partial pressure of oxygen | immediately after performing extracorporeal membrane oxygenation
  PO₂ is used to indicate the state of internal respiration.
Oxygen saturation | Before perform the extracorporeal membrane oxygenation
  SO₂ is used to indicate the state of internal respiration.
Oxygen saturation | immediately after performing extracorporeal membrane oxygenation
  SO₂ is used to indicate the state of internal respiration.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongwei Huang, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

REFERENCES:
- [Background] Masson R, Colas V, Parienti JJ, Lehoux P, Massetti M, Charbonneau P, Saulnier F, Daubin C. A comparison of survival with and without extracorporeal life support treatment for severe poisoning due to drug intoxication. Resuscitation. 2012 Nov;83(11):1413-7. doi: 10.1016/j.resuscitation.2012.03.028. Epub 2012 Mar 31. PMID 22469751
- [Background] Weiner L, Mazzeffi MA, Hines EQ, Gordon D, Herr DL, Kim HK. Clinical utility of venoarterial-extracorporeal membrane oxygenation (VA-ECMO) in patients with drug-induced cardiogenic shock: a retrospective study of the Extracorporeal Life Support Organizations' ECMO case registry. Clin Toxicol (Phila). 2020 Jul;58(7):705-710. doi: 10.1080/15563650.2019.1676896. Epub 2019 Oct 16. PMID 31617764
- [Background] Aso S, Matsui H, Fushimi K, Yasunaga H. In-hospital mortality and successful weaning from venoarterial extracorporeal membrane oxygenation: analysis of 5,263 patients using a national inpatient database in Japan. Crit Care. 2016 Apr 5;20:80. doi: 10.1186/s13054-016-1261-1. PMID 27044572
- [Background] Parker BM, Rao T, Matta A, Quitanna M, Reynolds HN, Stein DM, Haase D. Loperamide induced cardiac arrhythmia successfully supported with veno-arterial ECMO (VA-ECMO), molecular adsorbent recirculating system (MARS) and continuous renal replacement therapy (CRRT). Clin Toxicol (Phila). 2019 Nov;57(11):1118-1122. doi: 10.1080/15563650.2019.1580370. Epub 2019 Feb 26. PMID 30806091
- [Background] Mohan B, Gupta V, Ralhan S, Gupta D, Puri S, Mahajan R, Goyal A, Chhabra S, Tandon R, Aslam N, Wander GS, Singh B. Impact of extra-corporeal membrane oxygenation on outcome of aluminium phosphide poisoning complicated with myocardial dysfunction. Clin Toxicol (Phila). 2019 Nov;57(11):1095-1102. doi: 10.1080/15563650.2019.1584297. Epub 2019 Mar 11. PMID 30856020
- [Background] Tang X, Sun B, He H, Li H, Hu B, Qiu Z, Li J, Zhang C, Hou S, Tong Z, Dai H. Successful extracorporeal membrane oxygenation therapy as a bridge to sequential bilateral lung transplantation for a patient after severe paraquat poisoning. Clin Toxicol (Phila). 2015 Nov;53(9):908-13. doi: 10.3109/15563650.2015.1082183. Epub 2015 Aug 28. PMID 26314316
- See also: related information — http://www.elso.org/Home.aspx